CLINICAL TRIAL: NCT02898194
Title: Focus Groups to Determine Surrogates' Views Regarding Patient Preference Predictors
Brief Title: Focus Groups to Determine Surrogates Views Regarding Patient Preference Predictors
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 160168; 16-CC-0168
Record Dates: First submitted 2016-09-10; First posted 2016-09-13 (Estimated); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Normal Physiology
Keywords: Surrogate Decision-making; Health Care; Medical Decisions; End of Life Care; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Patient Surrogates: Any eligible participant who have acted as a surrogate medical decision-maker.

SUMMARY:
Background:

Some people cannot make medical treatment decisions on their own. The people who make decisions on their behalf are called medical surrogates. Sometimes surrogates cannot predict which treatment course the person or their loved ones would have chosen. The surrogates often become distressed because of making these decisions. Researchers think a tool called a Patient Preference Predictor (PPP) may be able to make the process easier. The PPP would predict what treatment the person would want. This is based on treatment preferences of similar people in a similar circumstance. Researchers want to interview surrogates to explore their views on the PPP.

Objective:

To explore surrogates views on incorporating a PPP into shared medical decision-making.

Eligibility:

People 18 years or older who:

Have acted as a surrogate medical decision-maker within the past 3 years. This includes decisions about

treatment, medication, hospice care, hospital admission, or discharge.

Are not pregnant

Design:

Participants will be screened by meeting with clinicians in person or by phone to discuss the study.

Participants will take part in a focus group. This is a small group of people discussing their thoughts and opinions. This will last for about 2 hours.

Participants will be served a light meal.

Participants will provide information about themselves and their views. They will talk about their past experiences making medical decisions for someone. They will discuss how they felt about these decisions.

The PPP will be explained to participants. They will give their views on it.

The research team will audio record the focus group and take notes.

Participants will fill out questionnaires.

DETAILED DESCRIPTION:
Current clinical practice relies on shared decision-making between clinicians and surrogates to make treatment decisions for patients who cannot decide on their own. This decision-making process is meant to promote medical care that accords with the patient s own preferences and values. However, empirical data suggest that this model faces two significant challenges. First, both surrogates and clinicians have trouble predicting which treatment course patients would have chosen. Second, given the nature of the decisions, surrogates often experience significant emotional distress as a result of making treatment decisions. To address these concerns it has been suggested that the shared decision-making process might be supplemented with a Patient Preference Predictor (PPP). A PPP would provide a prediction of which treatment a given patient would want based on the treatment preferences of similar patients in similar circumstances. The present study proposes to interview surrogates who have been involved in making decisions for an incapacitated patient to explore their perspectives on the PPP and how to incorporate it into medical decision-making for incapacitated patients..

ELIGIBILITY:
* INCLUSION CRITERIA:
* 18 years or older
* Experience making at least one medical decision on behalf of an incompetent patient within the past 3 years. A medical decision for the purposes of this study is defined as making a decision in a context in which there was more than 1 feasible or reasonable option.
* Ability to provide informed consent

EXCLUSION CRITERIA:

* Inability to speak, understand, or read English
* The patient on behalf of whom the individual acted as surrogate is deceased for less than two months.
* In the view of the referring clinician, participation in the study is deemed excessively burdensome.
* Candidate for study is pregnant
* Court appointed surrogate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any individual who acted as a surrogate decision maker for individuals undergoing any treatment.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Views of participants on PPP | Prior to, during, and immediately following the focus group session
  Level of acceptance regarding Patient Preference Predictor (PPP)

SECONDARY OUTCOMES:
Views of Participants on PPP as patients | Prior to, during, and immediately following the focus group
  Level of acceptance regarding PPP

CONTACTS AND LOCATIONS:
Overall Officials: David Wendler, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (2):
- United States (2):
  - St. Elizabeths Hospital, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, Bethesda, Maryland

REFERENCES:
- [Background] Shalowitz DI, Garrett-Mayer E, Wendler D. How should treatment decisions be made for incapacitated patients, and why? PLoS Med. 2007 Mar;4(3):e35. doi: 10.1371/journal.pmed.0040035. No abstract available. PMID 17388655
- [Background] Rid A, Wendler D. Use of a patient preference predictor to help make medical decisions for incapacitated patients. J Med Philos. 2014 Apr;39(2):104-29. doi: 10.1093/jmp/jhu001. Epub 2014 Feb 13. PMID 24526785
- [Background] Rid A, Wesley R, Pavlick M, Maynard S, Roth K, Wendler D. Patients' priorities for treatment decision making during periods of incapacity: quantitative survey. Palliat Support Care. 2015 Oct;13(5):1165-83. doi: 10.1017/S1478951514001096. Epub 2014 Oct 2. PMID 25273677
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-CC-0168.html